CLINICAL TRIAL: NCT00776750
Title: Influenza Vaccination in Hemodialysis Patients and Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML2394
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Hemodialysis; Renal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- influenza vaccination (Experimental): All participants received a standard dose of 0.5 ml commercially available trivalent split influenza vaccine (Vaxigrip®, Aventis Pasteur MSD) by intramuscular injection. The vaccine contained 15 μg hemagglutinin of each of the following influenza strains: A/ New Caledonia/20/99 (H1N1), A/ Panama/2007/99 (H3N2), and B/Shangdong/7/97, recommended by WHO as components of the influenza vaccine for the epidemic season 2003/2004.
  Interventions: Biological: trivalent split influenza vaccine

INTERVENTIONS:
Biological: trivalent split influenza vaccine — standard dose of 0.5 ml commercially available trivalent split influenza vaccine (Vaxigrip®, Aventis Pasteur MSD) by intramuscular injection

SUMMARY:
Disturbances of acquired immunity are considered to be responsible, at least partly, for the high infection rate and inadequate response to vaccinations observed in hemodialysis (HD) patients and renal transplant recipient (RTR). The present prospective trial aims at (a) evaluating the immunogenicity of a standard influenza vaccine in HD and RTR patients and (b) at identifying determinants of the immune response.

ELIGIBILITY:
Inclusion Criteria:

* maintenance hemodialysis patients or
* renal transplant recipients (beyond month 3 after transplantation)

Exclusion Criteria:

* patients with known allergy to chicken proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2003-09; Primary Completion 2004-05; Study Completion 2004-05

PRIMARY OUTCOMES:
Seroprotection rate, defined as the percentage of patients with an HI antibody titer ≥ 40,

SECONDARY OUTCOMES:
Seroresponse rate, defined as the percentage of patients with a fourfold rise in HI titer after vaccination; impact of booster vaccination on the immune response, and safety of influenza vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Vanrenterghem, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Scharpe J, Peetermans WE, Vanwalleghem J, Maes B, Bammens B, Claes K, Osterhaus AD, Vanrenterghem Y, Evenepoel P. Immunogenicity of a standard trivalent influenza vaccine in patients on long-term hemodialysis: an open-label trial. Am J Kidney Dis. 2009 Jul;54(1):77-85. doi: 10.1053/j.ajkd.2008.11.032. Epub 2009 Apr 1. PMID 19339089